CLINICAL TRIAL: NCT02310724
Title: Long-term Post-Intervention Follow-up of the TODAY Cohort (Treatment Options for Type 2 Diabetes in Youth and Adolescents)
Brief Title: TODAY2 Phase 2 Follow-up
Acronym: T2P2
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK61230-T2P2; U01DK061230 (NIH)
Record Dates: First submitted 2014-06-18; First posted 2014-12-08 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes
Keywords: youth onset type 2 diabetes; insulin sensitivity; beta cell function; macrovascular comorbidities; microvascular comorbidities
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine are collected annually and shipped to the study's Central Biospecimen Laboratory for analysis and storage.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TODAY cohort: All subjects randomized to the TODAY clinical trial are eligible to participate in T2P2. The study performs long-term observation only and administers no treatment, care, or management.
  Interventions: Other: TODAY cohort

INTERVENTIONS:
Other: TODAY cohort — This protocol is observation only and involves no intervention, care, treatment, or management.

SUMMARY:
The primary objective of T2P2 is to track the progression of T2D and related comorbidities and complications in the TODAY cohort as they transition to young adulthood. We hypothesize that:

* Youth-onset type 2 diabetes (T2D) will progress rapidly and result in high rates of diabetes-related medical complications and comorbidities.
* The rapid rate of progression is related to increased insulin resistance characteristic of puberty, worse β-cell function, degree of glycemic control, control of non-glycemic factors, and obesity itself.

ELIGIBILITY:
Inclusion Criteria:

* Participated in TODAY clinical trial.

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects randomized into the TODAY study are eligible to participate in T2P2. There are no additional inclusion or exclusions criteria for participation in T2P2.
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
diabetic retinopathy | year 4
  a microvascular complication determined by fundus photography
microalbuminuria | every 12 months
  a microvascular complication determined by urine albumin excretion >= 30 mg/day
overt diabetic nephropathy | every 12 months
  a microvascular complication determined by glomerular filtration rate < 70 mL/min/1.73m2
peripheral diabetic neuropathy | every 12 months
  a microvascular complication defined as the presence of Michigan Neuropathy Screening Instrument (MNSI) exam score >2 and <8 out of 10 appropriate responses to the Semmes-Weinstein monofilament (SW-MF) in either foot.
cardiac function | year 2
  a macrovascular (cardiovascular) risk indicator determined by echocardiogram
arterial stiffness | year 5
  a macrovascular (cardiovascular) risk indicator determined by pulse wave velocity
cardiovascular risk lipid values | every 12 months
  a macrovascular (cardiovascular) risk indicator determined by abnormal lipid value for LDL (>= 130 mg/dL) or triglycerides (>= 300 mg/dL)

SECONDARY OUTCOMES:
glycemic control | every 12 months
  determined by HbA1c (annual)
psychological disorder | every 12 months
  determined by scores on the following participant self-report standard surveys: (a) the Beck Depression Inventory II (BDI-II), (b) the Patient Health Questionnaire (PHQ) scales for somatic symptoms, anxiety, and alcohol use; participants are also interviewed about emotional or mental health problems involving referral, treatment, or hospitalization, and psychiatric diagnoses made by a non-study source that can be confirmed according to standard study criteria from acquired medical records are also recorded
body composition | every 12 months
  determined by body mass index (BMI) computed from physical measurements of height and weight
insulin sensitivity and beta cell function | participant years 6 and 9 from baseline
  determined by oral glucose tolerance test (at 6 and 9 years from randomization) to derive measures of insulin sensitivity (1/insulin0), insulin secretion (ΔC-peptide30-0/Δglucose30-0, Δinsulin30-0/Δglucose30-0 if not on insulin), and the oral disposition index (oDI = insulin sensitivity x insulin secretion)
eating disorder | every 12 months
  determined by score on participant self report questionnaire Eating Disorder Diagnostic Scale (EDDS)
health-related quality of life | every 12 months
  determined by score on the participant self report questionnaire Pediatric Quality of Life Inventory version 4.0 with age-specific versions for teen (13-18), young adult (19-25), and adult (≥26)
blood pressure | every 12 months
  determined by collection of blood pressure
sleep function | years 2-3
  determined by scores on standard questionnaires and in-lab polysomnogram
life stress | every 12 months
  determined by participant self report questionnaire based on the Yeaworth Adolescent Life Change Event Scale
healthcare usage | every 6 months
  determined by participant self report about visits, referrals, treatments, tests, and procedures related to healthcare

CONTACTS AND LOCATIONS:
Overall Officials: Philip S Zeitler, MD PhD, Study Chair — University of Colorado Denver Children's Hospital; Silva Arslanian, MD, Principal Investigator — University of Pittsburgh; Sonia Caprio, MD, Principal Investigator — Yale University; Jeanie B Tryggestad, MD, Principal Investigator — University of Oklahoma Health Science Center; Mitchell E Geffner, MD, Principal Investigator — Children's Hospital Los Angeles; Robin S Goland, MD, Principal Investigator — Columbia University Naomi Berrie Diabetes Center; Lorraine L Katz, MD, Principal Investigator — Children's Hospital of Philadelphia; Lori MB Laffel, MD, Principal Investigator — Joslin Diabetes Center; Jane L Lynch, MD, Principal Investigator — University of Texas Health Sciences Center at San Antonio; Siripoom V McKay, MD, Principal Investigator — Baylor College of Medicine; Rose Gubitosi-Klug, MD, Principal Investigator — Case Western Reserve University Rainbow Babies and Children's Hospital; David M Nathan, MD, Principal Investigator — Massachusetts General Hospital; Sherida E Tollefsen, MD, Principal Investigator — St. Louis University; Ruth S Weinstock, MD PhD, Principal Investigator — SUNY Upstate Medical Center; Neil H White, MD, Principal Investigator — Washington University School of Medicine
Locations (15):
- United States (15):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Colorado Denver Children's Hospital, Aurora, Colorado
  - Yale University School of Medicine Department of Pediatrics, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Columbia University Naomi Berrie Diabetes Center, New York, New York
  - SUNY Upstate New York University, Syracuse, New York
  - Case Western Reserve University Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The TODAY/TODAY2 Study Group engages in a number of methods to disseminate and share resources.
  * Findings are reported in manuscripts and presentations.
  * An active Ancillary Studies Committee reviews proposals to access the study cohort, the central database, and stored biospecimens.
  * Materials from the TODAY lifestyle intervention program and the standard diabetes education manual for adolescents developed by study experts are made available for public access on the website https://today.bsc.gwu.edu/web/today/home.
  * The study group adheres to the policies of the NIDDK Central Repositories to make data available to other scientific investigators. A TODAY2 de-identified database will be prepared and transferred along with excess stored biospecimens. Appropriate informed consent is required to transfer stored biospecimens.
  * TODAY establishes collaborative arrangements to work with other federally funded study groups.
Supporting Information: Study Protocol
Time Frame: Data will be prepared and provided to the NIDDK Data Repository in early 2022
Access Criteria: Currently with approval of the Ancillary Studies Committee and after 2022 as determined by the NIDDK Data Repository

REFERENCES:
- [Result] TODAY Study Group. Health Care Coverage and Glycemic Control in Young Adults With Youth-Onset Type 2 Diabetes: Results From the TODAY2 Study. Diabetes Care. 2020 Oct;43(10):2469-2477. doi: 10.2337/dc20-0760. Epub 2020 Aug 10. PMID 32778555
- [Result] TODAY Study Group. Longitudinal Changes in Cardiac Structure and Function From Adolescence to Young Adulthood in Participants With Type 2 Diabetes Mellitus: The TODAY Follow-Up Study. Circ Heart Fail. 2020 Jun;13(6):e006685. doi: 10.1161/CIRCHEARTFAILURE.119.006685. Epub 2020 Jun 5. PMID 32498621
- [Derived] Tryggestad JB, Drews KL, Mele L, Arslanian S, Chernausek SD, Escaname EN, Geffner M, Isganaitis E, Sprague J, Kelsey MM; TODAY Study Group. Impact of youth onset type 2 diabetes during pregnancy on microvascular and cardiac outcomes. Diabetes Res Clin Pract. 2023 Sep;203:110876. doi: 10.1016/j.diabres.2023.110876. Epub 2023 Aug 16. PMID 37595843
- [Derived] TODAY Study Group; Shah RD, Braffett BH, Tryggestad JB, Hughan KS, Dhaliwal R, Nadeau KJ, Levitt Katz LE, Gidding SS. Cardiovascular risk factor progression in adolescents and young adults with youth-onset type 2 diabetes. J Diabetes Complications. 2022 Mar;36(3):108123. doi: 10.1016/j.jdiacomp.2021.108123. Epub 2022 Jan 3. PMID 35123868
- [Derived] Trief PM, Uschner D, Tung M, Marcus MD, Rayas M, MacLeish S, Farrell R, Keady J, Chao L, Weinstock RS. Diabetes Distress in Young Adults With Youth-Onset Type 2 Diabetes: TODAY2 Study Results. Diabetes Care. 2022 Mar 1;45(3):529-537. doi: 10.2337/dc21-1689. PMID 35015056
- [Derived] TODAY Study Group; Bjornstad P, Drews KL, Caprio S, Gubitosi-Klug R, Nathan DM, Tesfaldet B, Tryggestad J, White NH, Zeitler P. Long-Term Complications in Youth-Onset Type 2 Diabetes. N Engl J Med. 2021 Jul 29;385(5):416-426. doi: 10.1056/NEJMoa2100165. PMID 34320286